CLINICAL TRIAL: NCT01470950
Title: Characterization of the Changes in the Signalling Pathways During Spinal Cord Injury-induced Skeletal Muscle Atrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinique Romande de Readaptation (Network)
Collaborators: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Principal Investigator, Bertrand LEGER, PhD, Scientific Collaborator, Clinique Romande de Readaptation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MMStudy
Record Dates: First submitted 2011-09-21; First posted 2011-11-11 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Spinal Cord Injuries; Muscle Atrophy
Keywords: Functional Electrical Stimulation; Signalling Pathways
MeSH Terms: conditions — Spinal Cord Injuries; Muscular Atrophy

ARMS (1):
- MotionMaker Training (Experimental): Device description: MotionMaker™ is a stationary robotic system for the active mobilization of the lower limbs. With its proprietary 'Closed-Loop' technology, it is a novel and exciting development that offers a truly interactive patient training system Training 3 times a week with MotionMaker device together with conventional treatment
  Interventions: Procedure: Motionmaker

INTERVENTIONS:
Procedure: Motionmaker — 3 times per week, FES Training on the Motionmaker device, for 6 months

SUMMARY:
Atrogin-1 and muscle RING finger-1 are skeletal muscle specific genes, with ubiquitin ligase activities, that are upregulated during muscle atrophy in mice. The Akt/GSK3 and Akt/mTOR pathways are involved in muscle hypertrophy in mice. Recent studies by the investigators team and others have demonstrated the implication of these signalling pathways in the control of muscle mass in humans. However no study has yet investigated the involvement of these systems in the early stages of spinal cord injury induced human skeletal muscle atrophy.

The investigators propose to investigate the level of expression of the different components of the ubiquitin-proteasome system together with the level of expression and activity of the Akt/mTOR and Akt/GSK3 signalling pathways after SCI in humans during the first months following the injury.

A second aim of this project is to assess if a novel apparatus of electrical stimulation which generate movements by closed-loop electrical muscle stimulation may improve strength and muscle mass in these patients.

The patients will be recruited jointly at the Clinique Romande de Réadaptation (CRR) in Sion and the Swiss paraplegic centre in Nottwil. They will be randomly divided into two groups, a first group of patients will undergo a conventional treatment of rehabilitation while a second set of patients will be treated using a brand new system of electro-stimulation called MotionMaker TM. Biopsies will be obtained in the first weeks after admission; two other biopsies will be taken respectively 3 and 6 months post-lesion.

Our results will provide an increased understanding of the molecular mechanisms contributing to skeletal muscle atrophy during the early stages following SCI and a characterization of the impact of endurance training in the no more voluntary innervated muscle. Moreover this study will also investigate the potential improvement in the rehabilitation process by using a new system of electro-stimulation.

DETAILED DESCRIPTION:
Measures:

For each group, the muscle biopsies will be divided into 3 samples which will be used for a) real-time PCR to quantify the gene expression of the different components of the ubiquitin-proteasome system (Atrogin-1, MuRF1, Nedd4, UBB and Psma) b) Western blotting, using anti-phospho-site specific antibodies to quantify the activities of the Akt/GSK3 and Akt/mTOR pathways and of their downstream regulators of protein synthesis, eIF2B, p70S6K and PHAS-1/4E-BP1and c) fiber type analysis to quantify the variation in MHC expression.

ELIGIBILITY:
Inclusion Criteria:

* acute, motor complete SCI
* lesion level C5-T12

Exclusion Criteria:

* diabetes type I
* pregnancy
* oral anti-coagulation
* osteosyntheses of the femur
* hepatitis B,C or D
* HIV

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Signaling pathways in human muscles after spinal cord injury | 6 months
  Molecular adaptations will be assessed from biopsies of the Vastus Lateralis muscle. Quantitative PCR method will allow to measure mRNA expression levels while proteins quantification will be performed by Western Blot analyses.

SECONDARY OUTCOMES:
Muscle strength | 6 months
  Improvement of muscle strenght
Spacity | 6 months
  Reduction of spasticity

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Léger, PhD, Principal Investigator — CRR Sion; Michael E Baumberger, MD, Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (2):
- Switzerland (2):
  - Swiss Paraplegic Centre, Nottwil, Canton of Lucerne
  - Clinique Romande de Réadaption, Sion, Valais